CLINICAL TRIAL: NCT07028359
Title: Sharp Health Companion App for Perioperative Education and Monitoring of Cataract Eye Surgery Patients Using CareKit Health Platform
Brief Title: Sharp Health Companion App for Cataract Surgery Preparation and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SHARP-CAT-RCT2022
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Cataract
Keywords: Cataract surgery; Mobile Health; Mhealth; Digital health; Medication adherence; Perioperative care; Older adults; Sharp health companion app; CareKit; iPhone
MeSH Terms: conditions — Cataract; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned 1:1 to printed instructions with phone reminders (Group 1) or to the Sharp Health Companion mobile app (Group 2), built using CareKit platform
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Group assignments were concealed from investigators, care teams, and outcomes assessors using a digital randomization app and unique study identifiers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Printed Instructions + Phone Reminders (Active Comparator): Participants in this arm received printed instructions for cataract surgery preparation and recovery, along with automated phone reminders. They used a printed checklist to track medication adherence. This group did not receive the Sharp Health Companion App.
  Interventions: Behavioral: Printed Instructions with Phone Reminders
- Group 2: Sharp Health Companion Mobile App Group (Experimental): Participants in this arm used the Sharp Health Companion App, a CareKit-based iPhone application, to receive digital pre- and postoperative instructions, medication reminders, and educational content. The app tracked medication adherence and surgical prep. Printed instructions were provided as backup.
  Interventions: Behavioral: Sharp Health Companion App (CareKit)

INTERVENTIONS:
Behavioral: Printed Instructions with Phone Reminders — Participants received paper-based instructions for perioperative care, including medication, fasting, and follow-up logistics. Automated phone calls were sent before surgery to reinforce preparation. Participants used a printed checklist to self-report eye drop adherence.
  Arms: Group 1: Printed Instructions + Phone Reminders
Behavioral: Sharp Health Companion App (CareKit) — The Sharp Health Companion App delivered interactive digital perioperative checklists, medication adherence prompts, COVID-19 protocol reminders, symptom tracking, and educational videos via iPhone. Participants logged their medication use in real time on the Sharp Health Companion App. Printed instructions were provided as a backup.
  Arms: Group 2: Sharp Health Companion Mobile App Group

SUMMARY:
This randomized controlled trial evaluated the effectiveness of the Sharp Health Companion App, a smartphone-based digital health tool, compared to standard printed instructions for supporting older adults undergoing cataract surgery. The study enrolled 200 patients aged 39-86 from a high-volume ophthalmology practice. Participants were randomly assigned to either a printed instructions group or a group using the mobile app built on Apple's CareKit platform. Outcomes included surgery cancellation rates, day-of-surgery delays, medication adherence (both subjective and objective), visual acuity, and patient satisfaction. The app significantly reduced same-day surgery delays and improved objective medication adherence. The study was completed between December 2022 and January 2024 and was approved by the Sharp HealthCare Institutional Review Board (IRB #2209803).

DETAILED DESCRIPTION:
This randomized controlled trial evaluated the effectiveness of the Sharp Health Companion App, a smartphone-based digital health tool, compared to standard printed instructions for supporting older adults undergoing cataract surgery. The study enrolled 200 patients aged 39-86 from a high-volume ophthalmology practice. Participants were randomly assigned to either a printed instructions group or a group using the mobile app built on Apple's open source CareKit platform. Outcomes included surgery cancellation rates, day-of-surgery delays, medication adherence (both subjective and objective), visual acuity, and patient satisfaction. The app significantly reduced same-day surgery delays and improved objective medication adherence. The study was completed between December 2022 and January 2024 and was approved by the Sharp HealthCare Institutional Review Board (IRB #2209803).

ELIGIBILITY:
Inclusion Criteria:

Scheduled for first-time cataract surgery at Sharp HealthCare Best-corrected visual acuity of 20/40 or worse Able to provide informed consent English-speaking For Group 2: possession of an iPhone and ability to use smartphone functions (e.g., Face ID or passcode)

Exclusion Criteria:

History of prior cataract surgery Significant cognitive, visual, or physical impairment preventing use of the app Inability to follow study procedures or complete follow-up Lack of access to compatible technology (Group 2 only)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Objective Medication Adherence Rate | 30 days post-surgery
  Percentage of patients whose surgery was delayed by two or more hours on the day of surgery due to noncompliance with preparation protocols (e.g., dietary, arrival time, or documentation errors).
Same-Day Cataract Surgery Delay Rate | Day of Surgery
  Percentage of patients whose surgery was delayed by two or more hours on the day of surgery due to noncompliance with preparation protocols (e.g., dietary, arrival time, or documentation errors).
Cataract Surgery Cancellation Rate | Day of schedule surgery
  Percentage of patients whose surgery was delayed by two or more hours on the day of surgery due to noncompliance with preparation protocols (e.g., dietary, arrival time, or documentation errors).

SECONDARY OUTCOMES:
Self-Reported Medication Adherence | 30 days post-surgery
  Percentage of patients whose surgery was delayed by two or more hours on the day of surgery due to noncompliance with preparation protocols (e.g., dietary, arrival time, or documentation errors).
Visual Acuity Outcome | Baseline to 30 days post-surgery
  Percentage of patients whose surgery was delayed by two or more hours on the day of surgery due to noncompliance with preparation protocols (e.g., dietary, arrival time, or documentation errors).
Patient Reported Surgical Experience Score | 30 days post-surgery
  Percentage of patients whose surgery was delayed by two or more hours on the day of surgery due to noncompliance with preparation protocols (e.g., dietary, arrival time, or documentation errors).
Postoperative custodial macular edema (CME) incidence | 30 days post-surgery
  Percentage of patients whose surgery was delayed by two or more hours on the day of surgery due to noncompliance with preparation protocols (e.g., dietary, arrival time, or documentation errors).
Postoperative Iritis Incidence | 30 days post-surgery
  Percentage of patients whose surgery was delayed by two or more hours on the day of surgery due to noncompliance with preparation protocols (e.g., dietary, arrival time, or documentation errors).

CONTACTS AND LOCATIONS:
Overall Officials: Tommy Korn, MD, Principal Investigator — Sharp Rees-Stealy Medical Group and Sharp HealthCare
Locations (1):
- Sharp Rees-Stealy Medical Group, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No